CLINICAL TRIAL: NCT04372082
Title: Efficacy of HYdroxychloroquine and DILtiazem-nIClosamide Combination for the Treatment of Non-severe Forms of SARS-CoV2 Infection in Patients With Co-morbidities: Multicenter, Randomized, Open-labeled Controlled Trial
Brief Title: Hydroxychloroquine or Diltiazem-Niclosamide for the Treatment of COVID-19
Acronym: HYdILIC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: evidence showed chloroquine is not effective against COVID-19
Sponsor: University Hospital, Lille (Other)
Collaborators: I-site University Lille North Europe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020_40; 2020-002188-72 (EudraCT Number)
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-04

CONDITIONS: Sars-CoV2
Keywords: Covid-19; Hydroxychloroquine; Dilitazem; Niclosamide
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care; Hydroxychloroquine; Niclosamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard of care (SOC) (Placebo Comparator)
  Interventions: Other: Standard of care (SOC)
- SOC + Hydroxychloroquine (Experimental)
  Interventions: Other: Standard of care (SOC); Drug: Hydroxychloroquine
- SOC + Diltiazem-Niclosamide (Experimental)
  Interventions: Other: Standard of care (SOC); Drug: Association of diltiazem and niclosamide

INTERVENTIONS:
Other: Standard of care (SOC) — SOC procedures including self-monitoring and medical follow-up of clinical signs and if necessary any other symptomatic treatment (paracetamol, antibiotics, steroids, oxygen…) during the whole study duration
Drug: Hydroxychloroquine — 200 mg x 3 per day during 10 days in addition to SOC
  Arms: SOC + Hydroxychloroquine
Drug: Association of diltiazem and niclosamide — niclosamide 500 mg x 4 at J1 then 500 mg x 2 per day + diltiazem 60 mg x 3 per day during 10 days in addition to SOC
  Arms: SOC + Diltiazem-Niclosamide

SUMMARY:
No optimal antiviral intervention has been yet validated to treat COVID-19 disease. Comorbidities, such as older age, obesity, diabetes, history of cardiovascular diseases are associated with poor prognosis.

This study aims to evaluate the efficacy of two experimental antiviral treatments, compared to standard of care (SOC), to prevent clinical worsening, hospitalization or death at day 14 in adults with documented SARS-CoV-2 infection, asymptomatic or with symptoms lasting less than 8 days, and associated comorbidities without any severity criteria of the disease at inclusion.

Participants will be randomized to receive SOC alone or SOC + hydroxychloroquine 200 mg three times a day during 10 days or SOC + association of niclosamide 2 g at J1 then 500 mg two times a day with diltiazem 60 mg three times a day during 10 days. Efficacy and tolerance of each treatments will be compared across the three treatment groups during the 28 days of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 test on nasopharyngeal swab
* Onset of symptoms <8 days prior to randomization
* NEWS score<4 AND no item ≥2
* At least one comorbidity among: age ≥ 70 years old, history of cardiac disease, diabetes, obesity, chronic kidney disease, chronic respiratory failure, immunosuppression, neoplasia, liver failure (stage ≥ Child-Pugh B)
* Fully able to understand the challenges of the trial
* Signed informed consent
* Covered by Health Insurance

Exclusion Criteria:

For all patients:

* Inability to decide to participate
* Pregnancy or breath feeding
* Hypersensitivity to any of the test drugs
* stage 4 or 5 chronic kidney disease (DFG <30 mL/min/1.73 m²)

For hydroxychloroquine arm:

* Long QT syndrome or QTc space >500 ms
* Treatment with piperazine, halofantrine, dasatinib, nilotinib, citalopram, escitalopram, hydroxyzine, domperidone
* Hepatic porphyria, retinopathy, known glucose-6-phosphate dehydrogenase deficiency,
* Heart rate <50/min
* hypokaliemia < 3.5 mmol/L

For diltiazem arm:

* Heart rate<40/min
* Sinus bradycardia, second- or third-degree atrioventricular block
* Left heart insufficiency with pulmonary stasis
* Treatment with dantrolene, pimozide, dihydroergotamine, ergotamine, nifedipine, ivabradine, esmolol, bêta-blockers (bisoprolol, carvedilol, metoprolol, nebivolol), fingolimod

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
death | At day 14
  Composite criteria
clinical worsening (composite criteria) | At day 14
  clinical worsening defined by at least one of the NEWS score item > 2 (temperature >39,1°C or<35°C, cardiac rate >111 or ≤40 bpm, respiratory rate > 21 or ≤8 cycles par minute, SaO2 ≤ 93% room air (if its measure is available),need of oxygen
Assisted-ventilation and/or hospitalization (composite criteria) | At day 14

SECONDARY OUTCOMES:
National Early Warning Score (NEWS) | at day 3, day 8, day 14 day 28
  clinical state as reflected by NEWS scoring, the clinical state of the patient regarding respiratory state as defined by the NEWS scoring system
cumulative incidence of hospitalizations | at day 14
cumulative incidence of the use of oxygen therapy, non-invasive ventilation or invasive ventilation ( composite criteria) | at day 14
Mortality | at day 14 and at day 28
  Number of patients death
cumulative incidence of viral shedding on SARS-CoV-2 rt-PCR on nasopharyngeal swab; | at day 3, day 8
adverse drug reactions | during study, up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Karine Faure, MD,PhD, Principal Investigator — University Hospital, Lille